CLINICAL TRIAL: NCT03541928
Title: Phase II Study Evaluating HSV-tk + Valacyclovir Gene Therapy in Combination With Androgen Deprivation Therapy, Brachytherapy, External Beam Radiotherapy, and Prostatectomy for High-Risk Prostate Cancer
Brief Title: Phase II High Risk Prostate Cancer Trial Using Gene & Androgen Deprivation Therapies, Radiotherapy, & Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, E. Brian Butler, Chair of Radiation Oncology Department, Houston Methodist Hospital, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00017515
Record Dates: First submitted 2018-05-10; First posted 2018-05-31 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: High-risk Prostate Cancer; Prostate Cancer
Keywords: gene therapy; untreated prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Genetic Therapy; Valacyclovir; bicalutamide; Leuprolide; Brachytherapy; Prostatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gene Therapy, ADT, RT, and Surgery (Experimental): The investigational gene therapy, ADV/HSV-tk, will be administered by injection into the prostate at 5 x 10[11] virus particles (1.25 x 10[11] virus particles per tumor quadrant in 4 quadrants) on day 0 and day 30.
  The recommended dose of Valacyclovir for this trial is 2 g orally t.i.d. for 14 days (day 1 to day 15 and days 31 to 45).
  The recommended dose for Bicalutamide therapy in combination with an LHRH analogue is one 50 mg tablet once daily (morning or evening).
  Leuprolide acetate 7.5mg depot injection will be injected monthly for a total of 2 months.
  Interventions: Drug: HSV-Tk; Drug: Valacyclovir; Drug: Bicalutamide; Drug: Leuprolide Acetate; Radiation: Brachytherapy, External beam radiotherapy; Procedure: Radical prostatectomy

INTERVENTIONS:
Drug: HSV-Tk — Injection of the HSV-tk gene therapy product in four quadrants of prostate to enhance the immune system via "bystander effect" in which cytotoxicity is conferred to non-transduced neighboring cells. In vivo bystander effects are likely due to a combination of host immunological responses and to gap junction-mediated transport of phosphorylated prodrug metabolites to surrounding cells.
  Other Names: Gene therapy; AdV-tk gene therapy; Herpes simplex virus thymidine kinase
Drug: Valacyclovir — The recommended dose for this trial is 2 g orally t.i.d. for 14 days (day 1 to day 15 and days 31 to 45). This dose has been calculated to give a similar AUC as 10 mg/kg of intravenous acyclovir administered every 8 hours. This is the same dose regimen used in a previous phase I clinical trial of ADV/HSV-tk plus acyclovir and topotecan in patients with recurrent ovarian cancer.
  Other Names: Valtrex
Drug: Bicalutamide — The recommended dose for Bicalutamide therapy in combination with an LHRH analogue is one 50 mg tablet once daily (morning or evening), with or without food. It is recommended that Bicalutamide be taken at the same time each day.
  The use of an oral antiandrogen with medical castration for the treatment of prostate cancer is referred to as combined androgen blockade (CAB). Compared with LHRH-agonist monotherapy, CAB with bicalutamide did not reduce overall QoL but provided an early improvement in QoL related to lower urinary tract symptoms and pain.
  Other Names: Casodex
Drug: Leuprolide Acetate — Leuprolide acetate 7.5 mg depot injection will be injected monthly for a total of 2 months.
  Other Names: Lupron
Radiation: Brachytherapy, External beam radiotherapy — On day 60, patient will undergo high dose rate (HDR) Brachytherapy. The patient will have 8-14 needle catheters inserted under ultrasound guidance. CT simulation and radiation treatment planning will be performed. The needle catheters will be connected to an HDR afterloader containing an Iridium 192 source. A single dose of 1250cGy will be delivered.
  Other Names: HDR; EBRT
Procedure: Radical prostatectomy — approximately 2-3 weeks after radiotherapy completion, patient will undergo radical retropubic prostatectomy. Use of laparoscopy or robotic assistance will be at the urologist's discretion. Lymph node dissection will be performed.
  Other Names: Prostatectomy

SUMMARY:
This is a prospective phase II study to assess the efficacy and toxicity of HSV-tk+ valacyclovir gene therapy in combination with androgen deprivation therapy, brachytherapy, external beam radiotherapy, and prostatectomy in previously untreated high-risk prostate cancer.

DETAILED DESCRIPTION:
This phase II study plans to assess efficacy and toxicity of HSV-tk+ valacyclovir gene therapy in combination with androgen deprivation therapy, brachytherapy, external beam radiotherapy, and prostatectomy in previously untreated high-risk prostate cancer patients.

Clinical response as evaluated by changes in serum PSA level and digital rectal examination as well as by histological alterations on re-biopsy and prostatectomy such as the presence of apoptosis, necrosis, tumor proliferation and immunologic response, will be assessed following HSV-tk + valacyclovir treatment. Blood samples will be taken for systemic immunological response, blood counts and liver functions tests. Toxicity will be graded by the Common Terminology Criteria for Adverse Events (CTCAE) and Radiation Therapy Oncology Group (RTOG) neuro-toxicity scores (See Appendices). Additionally, patients will be followed closely to assess nadir PSA, freedom from PSA-progression, and freedom from local and distant progression and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have biopsy proven adenocarcinoma of the prostate
* Patients in should have at least one or more of the following characteristics PSA>20, Gleason score 8-10, Primary Gleason pattern 5, >4 cores with Gleason 8-10, and Clinical stage T3a-T4.
* No prior surgical, hormonal, or radiotherapy prostate treatment.
* ECOG performance status 0-1
* No evidence of metastatic disease or other malignancy (except squamous or basal cell skin cancers.
* Patients must have PSA within 3 months of entry.
* Signed informed consent to participate in the study must be obtained from patients after they have been fully informed of the nature and potential risks of the study by the investigator (or his/her designee) with the aid of written information.
* Willing to provide biopsies as required by the study.
* Patients must have adequate baseline organ function as assessed by the following laboratory values before initiating the protocol:
* serum creatinine < 1.5 mg%
* T. bilirubin < 2.5 mg%, ALT and AST < 2x normal
* Pts > 100,000/mm3 , ANC> 1500 mm , Hgb> 10gm%
* Normal partial thromboplastin time (PTT) and Pro-Thrombin Time (PT)

Exclusion Criteria:

* Prior treatment with immunomodulatory therapy, immunotherapy, and/or gene vector therapy in the past 3 months.
* Any cytotoxic chemotherapy, RT, or immunotherapy or any investigational drug within 3 weeks of study treatment start.
* Evidence of metastatic disease
* Prostate volume >50cc
* Prior prostate surgery (hyperthermia, cryotherapy, etc.)
* Prior pelvic radiotherapy
* Prior androgen ablation hormonal therapy (except finasteride if discontinued > 3 mo. prior to enrollment)
* Patients on corticosteroids or any immunosuppressive drugs.
* History of liver disease, such as cirrhosis or active/chronic hepatitis B or C.
* History of or current alcohol misuse/abuse within the past 12 months.
* Known or suspected allergy or hypersensitivity to any component of the proposed regimen (gene vector/Valacyclovir).
* Inability to swallow food or any condition of the upper gastrointestinal tract that precludes administration of oral medications (Valacyclovir).
* No active malignancy except for non-melanoma skin cancer or in situ cervical cancer or treated cancer from which the patient has been continuously disease free for more than 5 years.
* Presence of active or suspected acute or chronic uncontrolled infection or history of immunocompromise, including a positive HIV test result.
* Patients < 18 years of age
* Unwilling or unable to comply with the study protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-02 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Biochemical control rate | 5-year biochemical disease free survival rate
  measured by PSA

SECONDARY OUTCOMES:
Overall survival rate | 5-year overall survival rate
  Measured at the end of the study
Pathologic complete response rate | After prostatectomy
  Measured by pathologic result of prostatectomy
Safety based on questionnaire and clinical adverse event monitoring | 5-year post treatment
  Measured by the Sexual Health Inventory for Men (SHIM), the International Prostate Symptoms Score (IPSS), and the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: E. Brian Butler, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Background] Zagars GK, Pollack A, Kavadi VS, von Eschenbach AC. Prostate-specific antigen and radiation therapy for clinically localized prostate cancer. Int J Radiat Oncol Biol Phys. 1995 May 15;32(2):293-306. doi: 10.1016/0360-3016(95)00077-C. PMID 7538498
- [Background] Al-Mamgani A, van Putten WL, van der Wielen GJ, Levendag PC, Incrocci L. Dose escalation and quality of life in patients with localized prostate cancer treated with radiotherapy: long-term results of the Dutch randomized dose-escalation trial (CKTO 96-10 trial). Int J Radiat Oncol Biol Phys. 2011 Mar 15;79(4):1004-12. doi: 10.1016/j.ijrobp.2009.12.039. Epub 2010 Apr 24. PMID 20421153
- [Background] Teh BS, Ayala G, Aguilar L, Mai WY, Timme TL, Vlachaki MT, Miles B, Kadmon D, Wheeler T, Caillouet J, Davis M, Carpenter LS, Lu HH, Chiu JK, Woo SY, Thompson T, Aguilar-Cordova E, Butler EB. Phase I-II trial evaluating combined intensity-modulated radiotherapy and in situ gene therapy with or without hormonal therapy in treatment of prostate cancer-interim report on PSA response and biopsy data. Int J Radiat Oncol Biol Phys. 2004 Apr 1;58(5):1520-9. doi: 10.1016/j.ijrobp.2003.09.083. PMID 15050332
- [Background] Teh BS, Aguilar-Cordova E, Vlachaki MT, Aguilar L, Mai WY, Caillouet J, Davis M, Miles B, Kadmon D, Ayala G, Lu HH, Chiu JK, Carpenter LS, Woo SY, Grant WH 3rd, Wheeler T, Thompson TC, Butler EB. Combining radiotherapy with gene therapy (from the bench to the bedside): a novel treatment strategy for prostate cancer. Oncologist. 2002;7(5):458-66. doi: 10.1634/theoncologist.7-5-458. PMID 12401909
- [Background] Yossepowitch O, Eggener SE, Bianco FJ Jr, Carver BS, Serio A, Scardino PT, Eastham JA. Radical prostatectomy for clinically localized, high risk prostate cancer: critical analysis of risk assessment methods. J Urol. 2007 Aug;178(2):493-9; discussion 499. doi: 10.1016/j.juro.2007.03.105. Epub 2007 Jun 11. PMID 17561152
- [Background] Freytag SO, Stricker H, Pegg J, Paielli D, Pradhan DG, Peabody J, DePeralta-Venturina M, Xia X, Brown S, Lu M, Kim JH. Phase I study of replication-competent adenovirus-mediated double-suicide gene therapy in combination with conventional-dose three-dimensional conformal radiation therapy for the treatment of newly diagnosed, intermediate- to high-risk prostate cancer. Cancer Res. 2003 Nov 1;63(21):7497-506. PMID 14612551
- [Background] Freytag SO, Movsas B, Aref I, Stricker H, Peabody J, Pegg J, Zhang Y, Barton KN, Brown SL, Lu M, Savera A, Kim JH. Phase I trial of replication-competent adenovirus-mediated suicide gene therapy combined with IMRT for prostate cancer. Mol Ther. 2007 May;15(5):1016-23. doi: 10.1038/mt.sj.6300120. Epub 2007 Mar 20. PMID 17375076
- [Background] Crook J, Ludgate C, Malone S, Perry G, Eapen L, Bowen J, Robertson S, Lockwood G. Final report of multicenter Canadian Phase III randomized trial of 3 versus 8 months of neoadjuvant androgen deprivation therapy before conventional-dose radiotherapy for clinically localized prostate cancer. Int J Radiat Oncol Biol Phys. 2009 Feb 1;73(2):327-33. doi: 10.1016/j.ijrobp.2008.04.075. Epub 2008 Aug 15. PMID 18707821
- [Background] Golden EB, Pellicciotta I, Demaria S, Barcellos-Hoff MH, Formenti SC. The convergence of radiation and immunogenic cell death signaling pathways. Front Oncol. 2012 Aug 7;2:88. doi: 10.3389/fonc.2012.00088. eCollection 2012. PMID 22891162
- [Background] Gulley JL, Arlen PM, Bastian A, Morin S, Marte J, Beetham P, Tsang KY, Yokokawa J, Hodge JW, Menard C, Camphausen K, Coleman CN, Sullivan F, Steinberg SM, Schlom J, Dahut W. Combining a recombinant cancer vaccine with standard definitive radiotherapy in patients with localized prostate cancer. Clin Cancer Res. 2005 May 1;11(9):3353-62. doi: 10.1158/1078-0432.CCR-04-2062. PMID 15867235
- [Background] Kroemer G, Galluzzi L, Kepp O, Zitvogel L. Immunogenic cell death in cancer therapy. Annu Rev Immunol. 2013;31:51-72. doi: 10.1146/annurev-immunol-032712-100008. Epub 2012 Nov 12. PMID 23157435